CLINICAL TRIAL: NCT00413218
Title: A Phase III, Double-blind, Randomized Study to Evaluate the Safety and Efficacy of BAL8557 Versus a Caspofungin Followed by Voriconazole Regimen in the Treatment of Candidemia and Other Invasive Candida Infections
Brief Title: Isavuconazole (BAL8557) in the Treatment of Candidemia and Other Invasive Candida Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9766-CL-0105; WSA-CS-008 (Other: Basilea Pharmaceutica Ltd); 2006-003951-18 (EudraCT Number); NCT00444366 (obsolete NCT alias)
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Candidiasis, Invasive; Candidemia; Mycoses
Keywords: Invasive Candida infections; BAL8557; ASP9766; Isavuconazole; Candidemia; Candidemia and other invasive candida infections; Phase III study
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia; Mycoses | interventions — isavuconazole; Caspofungin; Voriconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isavuconazole (ISA) (Experimental): Participants received 3 intravenous (IV) loading doses of 200 mg of isavuconazole on days 1 and 2, followed by an IV maintenance dose of 200 mg once daily from day 3 to day 56. On day 11 at the discretion of the investigator, non-neutropenic patients could switch from IV to oral therapy. Oral therapy consisted of 200 mg isavuconazole twice daily.
  Interventions: Drug: Isavuconazole
- Caspofungin (CAS)/Voriconazole (Active Comparator): Participants received 1 intravenous (IV) loading dose of 70 mg CAS on day 1, followed by an IV maintenance dose of 50 mg CAS from day 2 to day 56. On day 11 at the discretion of the investigator, non-neutropenic patients could switch from IV CAS to oral voriconazole comprising of a loading dose of 400 mg twice daily (BID) on the first day of oral therapy followed by standard dosing of 200 mg BID thereafter.
  Interventions: Drug: Caspofungin; Drug: Voriconazole

INTERVENTIONS:
Drug: Isavuconazole — Administered by intravenous infusion.
  Other Names: ASP9766; BAL8557
  Arms: Isavuconazole (ISA)
Drug: Caspofungin — Administered by intravenous infusion.
  Other Names: Cancidas
  Arms: Caspofungin (CAS)/Voriconazole
Drug: Voriconazole — Administered by intravenous infusion.
  Other Names: VFend
  Arms: Caspofungin (CAS)/Voriconazole

SUMMARY:
The purpose of the study is to compare the safety and efficacy of isavuconazole versus caspofungin followed by voriconazole in the treatment of candidemia and other invasive Candida infections.

DETAILED DESCRIPTION:
Candida infections, representing approximately 80% of all major systemic fungal infections, are the fourth most common cause of nosocomial bloodstream infections, with a mortality rate of 40%. Isavuconazole is not yet approved for the treatment of fungal infections. This study investigates the efficacy and safety of intravenous and oral isavuconazole. Patients are randomized to isavuconazole and the reference regimen. Patients with a positive blood- or deep tissue culture of candida fungi can be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with candidemia or with an invasive Candida infection
* Presence of fever, hypothermia or other appropriate local sign of infection
* Female patients must be non-lactating and at no risk of pregnancy

Exclusion Criteria:

* Patients with a sole diagnosis of mucocutaneous candidiasis, i.e. oropharyngeal, esophageal or genital candidiasis; or candidal lower urinary tract infection or Candida isolated solely from respiratory tract specimens
* Patients with candidemia who failed a previous antifungal therapy for the same infection
* Patients previously enrolled in a phase III study with isavuconazole
* Patients with a body weight <40kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2007-03-08 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2015-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (113):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Somero Research Corporation, Palm Desert, California
  - University of California Davis Health System, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - Idaho Falls Infectious Diseases PLLC, Idaho Falls, Idaho
  - Loyola University Hospital, Maywood, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mercury Street Medical Group, Butte, Montana
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Regional Infection Diseases Infusion Center Inc., Lima, Ohio
  - Temple University Health Sciences, Philadelphia, Pennsylvania
- Argentina (5):
  - Hospital Britanico de Buenos Aires, Capital Federal
  - Hospital General de Agudos Dr. Carlos G. Durand, Capital Federal
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma
  - Hospital General de Agudos Dr. Cosme Argerich, La Boca
- Australia (4):
  - Fremantle Hospital, Fremantle
  - Mater Adult Hospital, South Brisbane
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - ULB Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (10):
  - Hospital Felicio Rocho, Belo Horizonte
  - Hospital das Clinicas da Universidade Federal de Minas Gerai, Belo Horizonte
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Hospital das Clinicas da UFPR, Curitiba
  - Hospital Nossa Senhora das Gracas, Curitiba
  - Hospital Sao Lucas - PUCRS, Porto Alegre
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Universitario Clementino Fraga Filho, Rio de Janeiro
  - Hospital Universitario de Santa Maria, Santa Maria
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences - Henderson Site, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
- Chile (3):
  - Hospital Dr. Sotero del Rio, Puente Alto Santiago
  - Hospital del Salvador, Santiago
  - Hospital Dr. Hernan Henriquez Aravena, Temuco
- China (2):
  - West China Hospital of Sichuan University, Chengdu
  - Huashan Hospital Fudan University, Shanghai
- France (2):
  - Hôpital Hautepierre, Strasbourg
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (7):
  - Charite Campus Mitte, Berlin
  - Universitaet Koeln, Cologne
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum St. Georg, Leipzig
  - Universitaetsklinik Leipzig, Leipzig
  - Universitaetsklinikum Leipzig, Lübeck
  - Universitaetsklinikum Wuerzburg, Würzburg
- Hungary (2):
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
- India (10):
  - Kasturba Medical College and Hospital, Mangalore, Karna
  - Kasturba Medical College K. M. C. Hospital, Manipal, Karna
  - Amrita Institute Of Medical Science, Kochi, Kerala
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Mahara
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Metro Centre for Respiratory Diseases, Noida, National Capital Territory of Delhi
  - Apollo Hospitals Educational & Research Foundation, Chennai
  - Nizam's Institute of Medical Sciences, Hyderabad
  - AMRI Hospital, Kolkata
  - Christian Medical College & Hospital, Vellore Tamilnadu
- Israel (8):
  - Ha Emek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Universtiy Hospital - Ein Kerem, Jerusalem
  - Sapir Medical Center, Meir Hospital, Kfar Saba
  - Rabin MC, Petah
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky MC Ichilov Hospital Tel Aviv, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Ma, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ente Ospedaliero Ospedeli Galliera, Genova
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Ospedaliera di Verona-Ospedale Civile Maggiore, Verona
- Lebanon (2):
  - AUB Medical Center, Beirut
  - Rafik Hariri Uni Hospital, Beirut
- Malaysia (2):
  - Hospital Ampang, Ampang
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur
- Mexico (4):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Hospital Civil de Guadalajara Dr Juan I Menchaca, Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador, México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Urology Research Ltd, Hamilton
- Philippines (2):
  - De La Salle Health Sciences Institute- DLSUMC, Cavite City
  - Philippine General Hospital, Manila
- Russia (2):
  - S.I. Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - State Institution "Hematology Research Center" RAMS, Moscow
- Singapore (2):
  - Singapore General Hospital - Parent, Singapore
  - National Neuroscience Institute, Singapore
- Unitas Hospital, Lyttelton Centurion, South Africa
- Hospital del Mar, Barcelona, Spain
- Switzerland (2):
  - Hôpitaux Universitaires de Genève - HUG, Geneva
  - Universitaetsspital Zuerich, Zurich
- Thailand (6):
  - Siriraj Hospital, Bangkoknoi
  - Songklanagarind Hospital, Hat Yai
  - Maharat Nakhon Ratchasima Hospital, Muang
  - Srinagarind Hospital, Muang
  - Maharaj Nakorn Chiang Mai Hospital, Muang
  - Ramathibodi Hospital, Ratchathewi

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kullberg BJ, Viscoli C, Pappas PG, Vazquez J, Ostrosky-Zeichner L, Rotstein C, Sobel JD, Herbrecht R, Rahav G, Jaruratanasirikul S, Chetchotisakd P, Van Wijngaerden E, De Waele J, Lademacher C, Engelhardt M, Kovanda L, Croos-Dabrera R, Fredericks C, Thompson GR. Isavuconazole Versus Caspofungin in the Treatment of Candidemia and Other Invasive Candida Infections: The ACTIVE Trial. Clin Infect Dis. 2019 May 30;68(12):1981-1989. doi: 10.1093/cid/ciy827. PMID 30289478
- [Derived] McCormack PL. Isavuconazonium: first global approval. Drugs. 2015 May;75(7):817-22. doi: 10.1007/s40265-015-0398-6. PMID 25902926
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consenting male and female participants ≥ 18 with candidemia or an invasive Candida infection who had a positive blood or tissue culture obtained within 96 hours prior to randomization and meeting the inclusion/exclusion criteria were enrolled in the study.
Pre-assignment Details: Participants were stratified at randomization by geographical region and baseline neutropenic status.
Groups:
- Caspofungin (CAS)/Voriconazole: Participants received 1 intravenous (IV) loading dose of 70 mg CAS on day 1, followed by an IV maintenance dose of 50 mg CAS from day 2 to day 56. Participants with body weight > 80 kg received 70 mg CAS daily. On day 11 at the discretion of the investigator, non-neutropenic patients could switch from IV CAS to oral voriconazole comprising of a loading dose of 400 mg twice daily (BID) on the first day of oral therapy followed by standard dosing of 200 mg BID thereafter.
Period: Overall Study
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Started (Four hundred and fifty participants were randomized but 10 participants did not receive treatment.) | 223 | 227
Intent to Treat Population (ITT) (The ITT consisted of all randomized participants who received at least one dose of study drug.) | 221 | 219
Completed | 120 | 131
Not Completed | 103 | 96
Not completed — Randomized but didn't receive study drug | 2 | 8
Not completed — Death | 57 | 56
Not completed — Lost to Follow-up | 14 | 17
Not completed — Admin | 20 | 14
Not completed — Missing | 1 | 0
Not completed — Withdrawal by Subject | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole | Total
Number analyzed (Participants) | 221 | 219 | 440
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 58.0 (17.54) | 57.9 (16.88) | 58.0 (17.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 93 | 171
  Male | 143 | 126 | 269
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 150 | 144 | 294
  Black or African American | 11 | 7 | 18
  Asian | 56 | 64 | 120
  Other | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 19 | 45
  Not Hispanic or Latino | 187 | 195 | 382
  Missing | 8 | 5 | 13
Neutropenic Status: Presence or Absence of Neutropenia [Count of Participants; unit: Participants] — Participants were stratified by baseline neutropenic status (presence vs absence of neutropenia) defined as absolute neutrophil count (ANC) < 0.5 x 10^9/L [< 500/mm^3] for ≥ 10 days.
  Participants
    Presence | 25 | 24 | 49
    Absence | 196 | 195 | 391
Geographical Region [Count of Participants; unit: Participants] — Participants were stratified at randomization by geographical region. The region Western Europe includes countries in Western Europe (Belgium, France, Germany, Italy, Spain and Switzerland), Australia and New Zealand. Other regions include countries Argentina, Brazil, Chile, China, Hungary, India, Israel, Lebanon, Malaysia, Mexico, Philippines, South Africa, Russia, Singapore and Thailand.
  Participants
    North America | 38 | 33 | 71
    Western Europe | 54 | 56 | 110
    Other Regions | 129 | 130 | 259

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response of Success at the End of Intravenous Therapy (EOIV) as Determined by the Data Review Committee (DRC) Based on the Assessments of Clinical and Mycological Responses as Well as Alternative Systemic AFT Use
Description: A Data Review Committee (DRC) was established from independent experts in the field of fungal infections to determine diagnosis and outcomes independently of the investigators and sponsor. Success was defined as clinical response (complete or partial) and mycological response (eradication or presumed eradication) without the use of alternative systemic antifungal therapy (AFT) within 48 hours after the last dose of IV study medication.
Time Frame: End of Intravenous Treatment (EOIV) (Days 11-56)
Population: The ITT population consisted of all randomized participants who received at least one dose of study drug. The mITT population consisted of ITT participants who had documented invasive candidiasis or candidemia at baseline based on the assessment of the independent blinded DRC. Reporting arms included participants who switched to oral ISA and CAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants | 60.3 | 71.1
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; The adjusted treatment difference (ISA-CAS) was calculated by a stratified Cochran-Mantel-Haenszel (CMH) method with the strata of geographical region and baseline neutropenic status; Test type: Non-Inferiority — The lower bound of the 95% CI for the adjusted treatment difference was compared to the protocol prespecified noninferiority margin (NIM) value of -15%. If the lower bound were greater than -15%, isavuconazole would be declared as noninferior to caspofungin; Adjusted Treatment Difference (%) = -10.8, 95% CI 2-sided [-19.9 to -1.8] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

2. Secondary Outcome: Percentage of Participants With Overall Response of Success at Follow Up Visit 1 (FU1-2 Weeks After End of Treatment (EOT)) as Determined by the DRC Based on the Assessments of Clinical, Mycological Responses and Antifungal Therapy (AFT)
Description: A data review committee (DRC) was established from independent experts in the field of fungal infections to determine diagnosis and outcomes independently of the investigators and sponsor. Success was defined as clinical response (complete or partial) and mycological response (eradication or presumed eradication), without the use of alternative systemic AFT within 48 hours after the last dose of IV study medication.
Time Frame: End of Treatment (EOT) (Day 56) and FU1 (2 weeks after end of treatment)
Population: The mITT was the primary efficacy population and it consisted of ITT participants who had documented invasive candidiasis or candidemia at baseline based on the assessment of the independent blinded DRC. The isavuconazole and caspofungin group included participants who switched to oral isavuconazol and voriconazole.
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants | 54.8 | 57.2
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -2.7, 95% CI 2-sided [-12.2 to 6.8] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

3. Secondary Outcome: Percentage of Participants With Overall Response of Success at EOT and Follow Up Visit 2 (FU2) as Determined by the DRC Based on the Assessments of Clinical and Mycological Responses as Well as Alternative Systemic AFT Use at EOT and FU2
Description: A data review committee (DRC) was established from independent experts in the field of fungal infections to determine diagnosis and outcomes independently of the investigators and sponsor. Success was defined as clinical response (complete or partial) and mycological response (eradication or presumed eradication), without the use of alternative systemic antifungal therapy AFT within 48 hours after the last dose of IV study medication (for EOT analysis) or for continued treatment of the primary infection, or for recurrent or emergent infection by FU2, with no recurrent or emergent infection by FU2 (for FU2 analysis).
Time Frame: EOT (Day 56) and FU2 (6 weeks after end of treatment)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants
  EOT (Day 56) | 61.3 | 72.1
  FU2 (6 weeks after end of treatment) | 43.2 | 48.3
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at EOT (Day 56). The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference % = -10.9, 95% CI 2-sided [-19.9 to -1.9] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 2: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at FU2 (6 weeks after end of treatment). The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference % = -5.4, 95% CI 2-sided [-15.00 to 4.2] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

4. Secondary Outcome: Percentage of Participants With Clinical Response of Success at EOIV, EOT, FU1 and FU2 as Determined by the Data Review Committee (DRC)
Description: A data review committee (DRC) was established from independent experts in the field of fungal infections to determine diagnosis and outcomes independently of the investigators and sponsor. Success was defined as clinical response (complete or partial).
Time Frame: EOIV (Days 11-56), EOT (Day 56), FU1 (2 weeks after end of treatment) and FU2 (6 weeks after end of treatment)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants
  Success- End of Intravenous Treatment (EOIV) | 76.4 | 84.1
  Success- End of Treatment (EOT) | 76.4 | 84.6
  Success- Follow-up Visit 1 (FU1) | 67.8 | 67.7
  Success- Follow-up Visit 2 (FU2) | 52.8 | 58.2
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at EOIV (Days 11-56).The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -8.2, 95% CI 2-sided [-15.4 to -0.9] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 2: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted Treatment Difference (%) = -8.6, 95% CI 2-sided [-15.8 to -1.5] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 3: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at FU1 (2 weeks after end of treatment). The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -0.4, 95% CI 2-sided [-9.1 to 8.3] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 4: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at FU2 (6 weeks after end of treatment).The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -5.8, 95% CI 2-sided [-15.3 to 3.6] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

5. Secondary Outcome: Percentage of Participants With Mycological Response of Success at EOIV, EOT, FU1 and FU2 as Determined by the Data Review Committee (DRC)
Description: A data review committee (DRC) was established from independent experts in the field of fungal infections to determine diagnosis and outcomes independently of the investigators and sponsor. Success was defined as mycological response (Eradication or Presumed Eradication).
Time Frame: EOIV (Days 11-56), EOT (Day 56), FU1 (2 weeks after end of treatment) and FU2 (6 weeks after end of treatment)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants
  Success-EOIV | 70.9 | 85.6
  Success-EOT | 71.9 | 87.6
  Success-FU1 | 66.8 | 65.7
  Success-FU2 | 51.8 | 56.7
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at EOIV (Days 11-56). The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -14.9, 95% CI 2-sided [-22.7 to -7.0] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 2: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted Treatment Difference (%) = -15.9, 95% CI 2-sided [-23.5 to -8.4] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 3: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at FU1 (2 weeks after end of treatment).The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -0.7, 95% CI 2-sided [-8.1 to 9.6] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 4: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; [analysis description as in outcome 4, analysis 4]; Test type: Other; Adjusted Treatment Difference (%) = -5.2, 95% CI 2-sided [-14.7 to 4.3] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

6. Secondary Outcome: Percentage of Participants With Mycological Response of Success at Day 7 and EOT as Determined by The Investigator
Description: Success was defined as mycological response (eradication or presumed eradication).
Time Frame: Day 7 and EOT (Day 56)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants
  Day 7 | 61.3 | 72.1
  EOT | 72.9 | 81.1
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of adjusted treatment difference (ISA-CAS) at Day 7. The adjusted treatment difference (ISA-CAS) was calculated by a stratified CMH method with the strata of geographical region and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = -11.4, 95% CI 2-sided [-20.4 to -2.5] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 2: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted Treatment Difference (%) = -8.5, 95% CI 2-sided [-16.5 to -0.4] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

7. Secondary Outcome: Percentage of Participants With Clinical Response of Success at Day 7 and EOT as Determined by The Investigator
Description: Investigators defined clinical response as success if participants exhibited complete or partial clinical response after evaluation of clinical signs and symptoms.
Time Frame: Day 7 and EOT (Day 56)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Groups:
- Isavuconazole (ISA): Participants received 3 intravenous (IV) loading doses of 200 mg of isavuconazole on days 1 and 2, followed by an IV maintenance dose of 200 mg once daily from day 3 to day 56. On day 11 at the discretion of the investigator, non-neutropenic participants could switch from IV to oral therapy. Oral therapy consisted of 200 mg isavuconazole once daily.
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants
  Day 7 | 54.3 | 64.7
  EOT | 70.9 | 78.6
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; [analysis description as in outcome 6, analysis 1]; Test type: Other; Adjusted Treatment Difference (%) = -11.1, 95% CI 2-sided [-20.3 to -1.9] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation
Statistical Analysis 2: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; [analysis description as in outcome 3, analysis 1]; Test type: Other; Adjusted Treatment Difference (%) = -8.1, 95% CI 2-sided [-16.3 to 0.1] — The 95% CI for the adjusted treatment difference was calculated based on a normal approximation

8. Secondary Outcome: All-Cause Mortality (ACM) at Day 14 and Day 56
Description: All-cause mortality is represented as the percentage of participants who died on or before the analysis day. Participants who were lost to follow-up (i.e., unknown survival status) before the analysis day were counted as death. All-cause mortality was examined on Day 14 and Day 56.
Time Frame: Day 14 and Day 56
Population: The mITT was the primary efficacy population and it consisted of ITT participants who had documented invasive candidiasis or candidemia at baseline based on the assessment of the independent blinded DRC.
Measure: Number; unit: Percentage of Participants
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 199 | 201
Percentage of Participants
  Day 14 All-cause Mortality | 14.6 | 12.4
  Day 56 All-cause Mortality | 30.7 | 29.9
Statistical Analysis 1: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of all-cause mortality on Day 14. Adjusted treatment difference (Isavuconazole-Caspofungin) is calculated by a stratified CMH method with the strata of geographical regions, and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = 2.5, 95% CI 2-sided [-3.8 to 8.9]
Statistical Analysis 2: Comparison: Isavuconazole (ISA) vs Caspofungin (CAS)/Voriconazole; Statistical analysis of all-cause mortality on Day 56. Adjusted treatment difference (Isavuconazole-Caspofungin) is calculated by a stratified CMH method with the strata of geographical regions, and baseline neutropenic status; Test type: Other; Adjusted Treatment Difference (%) = 1.4, 95% CI 2-sided [-7.1 to 10.0]

9. Secondary Outcome: Time to First Confirmed Negative Culture
Description: The first confirmed negative blood culture was defined as the first negative blood culture on or after first dose followed by a second negative blood culture at least 24 hours apart without any positive blood cultures in between. A participant without a confirmed negative blood culture was censored on the participant's last visit day. This endpoint was analyzed for mITT participants with candidemia only using the Kaplan-Meier method. Only participants with at least one positive blood culture on or prior to first dose and the culture not resolved prior to first dose were included in this analysis
Time Frame: Day 1 up to FU1 (2 weeks after EOT (Day 56))
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
Number analyzed (Participants) | 120 | 119
Days | 4.0 [3.0 to 6.0] | 3.0 [3.0 to 4.0]

ADVERSE EVENTS:
Time Frame: Day 1 to FU2 (6 weeks after EOT (Day 56))
Description: Treatment-emergent adverse events (TEAE) are AEs which started after the first use of study drug until FU2, and are based on the Safety Analysis Set (SAF) population. The SAF consisted of all participants who received at least one dose of study drug. SAF data were analyzed according to the first dose of study drug participants received even if it was different from what they were randomized to. One participant randomized to ISA received CAS on Day 1 and was included in CAS group for safety.
Groups:
- Isavuconazole (ISA): Participants received 3 intravenous (IV) loading doses of 200 mg of isavuconazole on days 1 and 2, followed by an IV maintenance dose of 200 mg once daily from day 3 to day 56. On day 11 at the discretion of the investigator, non-neutropenic patients could switch from IV to oral therapy. Oral therapy consisted of 200 mg isavuconazole once daily.
Arm/Group | Isavuconazole (ISA) | Caspofungin (CAS)/Voriconazole
All-Cause Mortality (participants affected / at risk) | 55/220 | 55/220
Serious Adverse Events (participants affected / at risk) | 112/220 | 106/220
Other Adverse Events (participants affected / at risk) | 162/220 | 167/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isavuconazole (ISA) (N=220) | Caspofungin (CAS)/Voriconazole (N=220)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (6) | 6 (6)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 5 (5) | 7 (7)
Necrosis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 2 (3) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Bacterial sepsis (Infections and infestations) | 3 (3) | 4 (4)
Candida endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebral aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 2 (2) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 16 (16) | 9 (9)
Septic shock (Infections and infestations) | 19 (19) | 11 (12)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Donor site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 2 (2) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 3 (3) | 0 (0)
Diabetic complication (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's disease refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basilar artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1)
Nephrectasia (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 10 (10) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 8 (8)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 2 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isavuconazole (ISA) (N=220) | Caspofungin (CAS)/Voriconazole (N=220)
Anaemia (Blood and lymphatic system disorders) | 13 (14) | 18 (21)
Tachycardia (Cardiac disorders) | 18 (20) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 16 (17) | 20 (23)
Constipation (Gastrointestinal disorders) | 32 (34) | 24 (31)
Diarrhoea (Gastrointestinal disorders) | 33 (37) | 41 (49)
Nausea (Gastrointestinal disorders) | 21 (28) | 30 (37)
Vomiting (Gastrointestinal disorders) | 33 (44) | 37 (49)
Chills (General disorders) | 11 (15) | 6 (6)
Oedema peripheral (General disorders) | 15 (17) | 16 (17)
Pyrexia (General disorders) | 38 (56) | 41 (73)
Bacteraemia (Infections and infestations) | 11 (12) | 9 (9)
Staphylococcal bacteraemia (Infections and infestations) | 13 (13) | 9 (10)
Urinary tract infection bacterial (Infections and infestations) | 7 (7) | 12 (12)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 11 (12)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 11 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (19) | 18 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 41 (49) | 44 (50)
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 (22) | 29 (31)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (12) | 14 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 15 (15) | 9 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (15) | 6 (6)
Agitation (Psychiatric disorders) | 5 (5) | 13 (15)
Anxiety (Psychiatric disorders) | 11 (11) | 7 (8)
Insomnia (Psychiatric disorders) | 12 (13) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 13 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 14 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 14 (15) | 10 (19)
Hypertension (Vascular disorders) | 9 (9) | 12 (13)
Hypotension (Vascular disorders) | 22 (30) | 27 (29)
Phlebitis (Vascular disorders) | 14 (14) | 15 (20)

LIMITATIONS AND CAVEATS:
Enrollment in the clinical study was suspended in January 2009 pending further characterization of newly identified impurities. After successful completion of the studies, regulatory notifications and transfer of sponsorship from Basilea to Astellas,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the Sponsor at least 1 month prior to the submission of any such information to an editorial board or scientific review committee. This allows the Sponsor to protect proprietary information and to provide comments based on information from other studies that may not yet be available to the investigator.